CLINICAL TRIAL: NCT06318780
Title: Concordance of Three Imaging Methods by Dynamic CT, Contrast Ultrasound and CT Angiography in the Characterization of Endoleaks in Patients With an Aortic Endoprosthesis
Acronym: LEAKDYN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2023_843_0171
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Aortic Diseases
Keywords: EVAR; d-CTA; CEUS
MeSH Terms: conditions — Aortic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: three-phase CT angiography — three-phase CT angiography
Other: CEUS ultrasound — CEUS ultrasound

SUMMARY:
Among patients who have undergone EVAR, there is a significant risk of 20-50% endoleak. These endoleaks often require secondary interventions to reduce the risk of expansion or rupture. Currently, three-phase CT angiography and CEUS ultrasound are recommended in the post-operative monitoring of EVAR but these remain limited in characterizing the type and source of endoleak. In this study the investigators will study the interest of d-CTA for a better detection and characterization of endoleaks.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age and older,
* Patients who have received EVAR ,
* Detection of endoleak and/or with an aneurysmal sac enlargement greater than or equal to 5 mm over 6 months.

Exclusion Criteria:

* Minor patients,
* absence of endoleak and growth of the aneurysmal sac (greater than or equal to 5 mm over 6 months),
* patient under guardianship, curators, safeguard of justice,
* patient deprived of liberty,
* pregnant woman
* Patient who does not benefit from a social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Endoleak classification using the CT angiography | 5 years
  Endoleak classification using the CT angiography
Variation of Endoleak classification between CEUS ultrasound and the CT angiography | 5 years
  Variation of Endoleak classification between CEUS ultrasound and the CT angiography

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No